CLINICAL TRIAL: NCT07368920
Title: A Prospective, Open-Label, Single-Arm, Self-Controlled Study of Transcutaneous Electrical Nerve Stimulation (TENS) for Adult Low Back Pain
Brief Title: Transcutaneous Electrical Nerve Stimulation (TENS) for the Treatment of Low Back Pain (LBP) in Adults
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xijing Hospital (Other)
Responsible Party: Principal Investigator, Bo Gao, MD, principal investigator, Xijing Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KY20252517
Record Dates: First submitted 2026-01-20; First posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Low Back Pain; Paraspinal Muscles; CLBP - Chronic Low Back Pain
Keywords: Low back pain; Transcutaneous electrical stimulation; Self-controlled clinical trial
MeSH Terms: conditions — Low Back Pain | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Intervention Model Description: This is a prospective, open-label, single-arm, self-controlled study. All enrolled participants will receive transcutaneous electrical stimulation (TENS) with a fixed treatment course of 5 sessions per week for 4 consecutive weeks, with stimulation parameters adjusted within a safe range based on individual tolerance. There is no parallel comparator group; each participant serves as their own control. Outcomes will be assessed at baseline and at Weeks 1, 2, 3, and 4 after treatment initiation, and adverse events/complications will be recorded throughout the study period.
Masking Description: This is an open-label study with no masking. Participants, care providers, investigators, and outcome assessors are all aware of the intervention assignment, as all participants receive the same TENS intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Transcutaneous Electrical Stimulation (TENS)） (Experimental): All enrolled participants in this arm will receive transcutaneous electrical nerve stimulation (TENS) therapy 5 times per week for 4 consecutive weeks. Treatment will be delivered according to a standardized protocol, with stimulation intensity adjusted within a safe range based on individual tolerance. Outcomes will be assessed at baseline and weekly during the 4-week treatment period, and adverse events will be recorded.
  Interventions: Device: Transcutaneous Electrical Nerve Stimulation (TENS)

INTERVENTIONS:
Device: Transcutaneous Electrical Nerve Stimulation (TENS) — TENS will be delivered via surface electrodes placed bilaterally around the area of maximal low back pain. Each session will last 20-30 minutes, administered 5 times per week for 4 weeks. Stimulation intensity will be titrated to a strong but comfortable sensation without pain, and parameters may be adjusted based on participant tolerance. Safety will be monitored throughout treatment and follow-up.

SUMMARY:
The goal of this clinical trial is to assess the effects and safety of transcutaneous electrical nerve stimulation (TENS) in adults with myofascial low back pain. Eligible participants will receive TENS treatment 5 times per week for 4 weeks. Pain intensity and functional outcomes will be assessed at baseline and weekly during the 4-week treatment period, and adverse events will be recorded.

DETAILED DESCRIPTION:
This study is a prospective, open-label, single-arm, self-controlled clinical trial conducted at the Department of Orthopaedics, Xijing Hospital. A total of 40 adult participants with myofascial low back pain will be recruited according to predefined inclusion and exclusion criteria and enrolled after providing written informed consent.

All enrolled participants will receive transcutaneous electrical stimulation (TENS) therapy with a treatment schedule of 5 sessions per week for 4 consecutive weeks. The stimulation parameters and single-session duration will be set within a safe range and may be adjusted according to individual tolerance.

Outcome assessments will be performed at baseline (Day 0, before intervention) and at Weeks 1, 2, 3, and 4 after treatment initiation. Pain intensity will be evaluated using the Visual Analog Scale (VAS; 0-10). Secondary outcomes include the Oswestry Disability Index (ODI), Japanese Orthopaedic Association (JOA) score, and the Short Form-36 (SF-36) to assess functional status and quality of life.

Safety will be monitored throughout the study, with adverse events and complications recorded during the study period and follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 18-65 years
2. Diagnosis consistent with myofascial low back pain (localized low back pain with a palpable taut band; referred pain and/or sensory changes near a specific trigger point; an identifiable tender spot within the taut band; mild muscle weakness and/or some limitation of joint range of motion)
3. Mild pain intensity at baseline (VAS < 4 on a 0-10 scale)
4. Symptom duration > 1 month
5. Able to understand the study procedures and demonstrate good compliance/cooperation
6. Written informed consent provided

Exclusion Criteria:

1. Low back pain due to other causes, including but not limited to lumbar disc herniation, lumbar spinal stenosis, ankylosing spondylitis, spinal tumor, spinal tuberculosis, or spinal infection
2. Received physical therapy, interventional procedures, or medication treatment within 4 weeks prior to enrollment that may affect pain or function assessment
3. Systemic disease or organ dysfunction
4. Skin/soft tissue breakdown or infection at/near the planned treatment area
5. Use of sedative medications or opioid analgesics within 6 months prior to enrollment, or currently receiving other treatments that may affect study outcomes
6. Severe psychiatric disorder or inability to cooperate with study procedures
7. Pregnant or breastfeeding women

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2029-01-01 (Estimated); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
Pain Intensity Assessed by Visual Analog Scale (VAS) Score | Baseline (Day 0, pre-intervention), Week 1, Week2, Week3 and Week 4 after treatment initiation (end of treatment at Week 4).
  Pain intensity will be assessed using the Visual Analog Scale (VAS), a validated tool with a score range from 0 to 10 points. A score of 0 represents no pain, and a score of 10 represents the most severe pain imaginable. This outcome measure evaluates changes in pain intensity in adults with chronic low back pain (cLBP) following treatment with oral sodium aescinate tablets.

SECONDARY OUTCOMES:
Disability Severity Assessed by Oswestry Disability Index (ODI) Score | Baseline (Day 0, pre-intervention), Week 1, Week2, Week3 and Week 4 after treatment initiation (end of treatment at Week 4).
  Disability related to low back pain will be assessed using the Oswestry Disability Index (ODI), a widely used questionnaire with a total score range of 0 to 50 points. Higher scores indicate greater disability in activities of daily living. This outcome measure evaluates changes in functional disability in cLBP patients after treatment.
Lumbar Functional Status Assessed by Japanese Orthopaedic Association (JOA) Score | Baseline (Day 0, pre-intervention), Week 1, Week2, Week3 and Week 4 after treatment initiation (end of treatment at Week 4).
  Lumbar spine function will be evaluated using the Japanese Orthopaedic Association (JOA) score, which ranges from 0 to 29 points. Lower scores indicate more severe functional impairment. This outcome measure assesses changes in lumbar spine function following treatment.
Health-Related Quality of Life Assessed by SF-36 Total Score | Baseline (Day 0, pre-intervention), Week 1, Week2, Week3 and Week 4 after treatment initiation (end of treatment at Week 4).
  Health-related quality of life will be assessed using the 36-Item Short Form Health Survey (SF-36). The total score ranges from 0 to 100 points, with higher scores indicating better overall health status. This outcome measure evaluates changes in overall quality of life in cLBP patients following treatment.
Lumbar Paraspinal Muscle Cross-Sectional Area Assessed by MRI | Baseline (Day 0, pre-intervention) and Week 4 after the start of treatment
  Lumbar MRI will be used to measure the cross-sectional area of paraspinal muscles as an objective indicator of muscle mass. This outcome measure evaluates changes in paraspinal muscle size following treatment with sodium aescinate tablets.
Lumbar Paraspinal Muscle Fat Infiltration Rate Assessed by MRI | Baseline (Day 0, pre-intervention) and Week 4 after the start of treatment
  Lumbar MRI will be used to assess the fat infiltration rate of paraspinal muscles as an indicator of muscle quality. This outcome measure evaluates changes in paraspinal muscle composition following treatment.

OTHER OUTCOMES:
Incidence of Adverse Events During Treatment | Within 4 weeks after the start of treatment (during the 4-week treatment period).
  All adverse events (AEs) occurring during the 4-week TENS treatment period will be recorded. For each AE, the event type, severity, onset and duration, action taken (if any), outcome, and the investigator-assessed relationship to the TENS intervention/device will be documented to evaluate safety and tolerability.

CONTACTS AND LOCATIONS:
Locations (1):
- Xjing hospital, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No